CLINICAL TRIAL: NCT01379820
Title: Use of Orotracheal CPAP ( Gregory System) for Treatment of Respiratory Failure in Newborns
Brief Title: Use of Orotracheal Continuous Positive Airway Pressure (CPAP) in Newborns With Respiratory Failure
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Angeles del Pedregal (Other)
Responsible Party: Head , Neonatology Department, Hospital Angeles del Pedregal.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01/2008
Record Dates: First submitted 2011-06-22; First posted 2011-06-23 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Neonatal Respiratory Failure
Keywords: NEONATAL RESPIRATORY FAILURE; OROTRACHEAL cpap; NASAL cpap; MECHANICAL VENTILATION; PNEUMOTHORAX; COMPENSATION BAG
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: OROTRACHEAL cpap WITH COMPENSATION BAG ( GREGORY CPAP) — USE OF OROTRACHEAL CPAP FOR RESPIRATORY DISTRESS SYNDROME IN NEWBORNS .

SUMMARY:
Nasal CPAP is a excellent ventilation modality for newborns, but the incidence of pneumothorax is high (65.% - 9%) our hypothesis is when the baby open the mouth or crie the pressure in the airway is variable, the investigators evaluate a closed system with a intubated baby with a orotracheal system but with a elastic reservoir , the reservoir distend and the pressure in the airway is constant ,with this system the investigators protect the lungs for damage . The investigators want compare the use of nasal CPAP, mechanical ventilation and orotracheal CPAP with a compensation bag (gregory system) in newborns with respiratory failure .

DETAILED DESCRIPTION:
Recent advances in the intensive care of the newborns are closely related to the evolution in the management of the respiratory distress syndrome (RDS) frequently associated with lung immaturity specially in the premature infant as well as with various pathological conditions in the mature lung of the full- term baby. The methods of ventilatory assistance to treat these conditions vary from continuous positive airway pressure (CPAP) to conventional mechanical ventilation and/or high frequency ventilation. It is reasonable to assume that the type of ventilatory assistance provided to these infants should be graded in accordance to the severity of the respiratory problem (1) therefore the mode of respiratory support should be one which while providing adequate ventilatory assistance will result in minimal volu or barotrauma.

Currently the investigators know that the best ventilatory technique is one that stabilizes Po2, Pco2 and Ph and avoids volu and barotrauma, diminishes the possibility of pulmonary injury and shortens the time spent in the hospital.

It has been demonstrated that with the use of CPAP the need for mechanical ventilation is less and that the possibility of pulmonary injury and the length of hospital stay are shortened (1 ) ( 2). The need to use mechanical ventilation increases when gestational age is marginal or in the presence of severe pulmonary pathology that causes increased respiratory problems which in turn enhances the possibility of increase the alveolar oxygen tension gradient (A-a DO2) to more then 180mmHg and to cause the presence of a more severe hyaline membrane syndrome as evidenced by sequential chest X rays (8). This also will limit the need for early nasal continuous airway pressure (ENCPAP). Other limiting factors could be pressure changes due to physiological events such as cry, mouth open or close, cough or hippus. In the past use CPAP generated by the ventilator administered via an endotracheal cannula ; however this method of ventilation has been abandoned due to the high risk of barotrauma due to the surges of pression in a closed, rigid, system that could eventually generate an increased resistance due to the disparity between the caliber of the endotracheal tube and that of the trachea (9). This increased resistance was for a long time considered to be a great limiting risk for the use of orotracheal CPAP particularly in premature infants.

According with the severity of the disease, the best results have been obtained with the use of low pressure, high pulmonary volumes such as those provided by high frequency oscillatory ventilation (HFOV) or conventional ventilation with a high positive end expiration pressure (PEEP) (1).

The investigators want determinate the rate of pneumothorax , use of oxygen at 36 weeks of gestational age , failure to treatment, mortality , infection rate an other complications with the 3 methods for assisted ventilation.

The concept of The Compensation Bag (accessory lung):

This concept is based on the gregory original work in 1972 (3) , the investigators postulate that the air pressure in a closed airway circuit always tries to find a way to escape, in this situation, the weakest point in this close circuit is the alveolus, therefore any variation in pressure will be directly reflected in the intrinsic alveolar pressure, that is, if there is a fall in the circuit pressure the intra-alveolar pressure will fall, causing in turn a decrease in the alveolar oxygen tension gradient which will cause a collapse of the alveolar sac. On the other hand an increase in the pressure of the airway circuit will augment the intra-alveolar pressure, distending the sac, causing inflammatory changes on its wall and eventually rupturing it occasioning air leakage and on the long run giving raise to pathological sequels such as bronchopulmonary dysplasia.

The compensation bag is fitted with a distensible mechanical valve which is interposed in the closed circuit, so that in case of an increase in pressure the distention point will be the bag and not the alveolus. Also in case of a decreased in pressure the point of collapse is the bag therefore preventing a collapse of the alveolar sac, this allows to maintain an optimally expanded alveolus without the risk of over distention or collapse. At the same time the pulmonary resistance occasioned by the endotracheal tube is regulated within the circuit thus improving the performance of the mechanical ventilation through a better alveolar expansion and a more adequate alveolar oxygen tension, avoiding sudden pressure variations but maintaining the benefit of conventional CPAP keeping a constant alveolar volume regardless of any physiological event.

In 1972 the Gregory work report excellent evolution with the use of a anesthestic bag for ventilation in newborns, in 2009 , the investigators reported a small study with a modified gregory system with excellent evolution . (4) in this work the investigators want report the use of this system in more babies .

ELIGIBILITY:
Inclusion Criteria:

* newborns with respiratory disease preterm less 32 week of gestational age.

Exclusion Criteria:

* newborns without respiratory disease or 33 week of gestational age or more.

Min Age: 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
mortality. pneumothorax , oxygen at 36 weeks of gestational age | at 36 weeks of gestational age
  we compare mortality. pneumothorax , oxygen at 36 weeks of gestational age in all the groups , mechanical ventilation , Nasal CPAP and orotracheal CPAP

SECONDARY OUTCOMES:
infections rate, failure to treatment , other complications. | 36 weeks of gestational age
  we compare infections rate, failure to treatment , other complications. in all the groups